CLINICAL TRIAL: NCT02659982
Title: Study Protocol for Evaluation of EarlySense Home Care Tele-monitoring Device - A Contact-Free System for Measuring Heart Rate, Respiratory Rate and Motion For Early Detection of Deterioration For Cardiac Patients at Home
Brief Title: Evaluation of EarlySense Home Care Tele-monitoring Device -For Early Detection of Deterioration For Cardiac Patients at Home
Status: Completed | Type: Observational
Sponsor: EarlySense Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-H-003-2013
Record Dates: First submitted 2015-12-28; First posted 2016-01-21 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2016-09

CONDITIONS: Post Cardiac Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study is to evaluate the relevance of the information as provided by the EarlySense Home care Tele-monitoring system can provide relevant flagging information for clinicians to identify the patients at higher risk to proactively assess patients' condition

DETAILED DESCRIPTION:
Study objectives include:

1. Assess if and to what extent the flags provided by EarlySense Home care tele-monitoring provides relevant clinical information that can help case managers / nurses of home care agency to detect patients who need further assessment and perhaps early intervention to minimize hospitalization (re-admission to hospital).
2. Use data to further optimize a decision algorithm utilizing changes in physiological data over time (i.e., hours to days) which may identify patients at higher risk for poor outcomes (flagging algorithm).
3. Assess the acceptability of the EarlySense Home care device by clinicians
4. Assess the acceptability of the EarlySense Home care device by patients at home and their families, in their own home as determined by a provided questioner

ELIGIBILITY:
Inclusion Criteria:

* Age 21 and up
* Any patient hosted in Shelev with geographically resident over 50 km from Sheba Medical Center/ Shelev
* Patients agrees to sign the consent form and comply with study protocol.

Exclusion Criteria:

* Patients do not agree to sign the consent form
* Planned readmission within 30 days of discharge from hospital
* Going home to hospice care.
* Patients with cognitive constraints or disabilities

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post Cardiac Surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
To evaluate if Alerts and Flags generated by the EarlySense Home Care System, could have potentially prevented readmission to hospitals, and providing better care at home, for post cardiac surgery patients | 30 days
  Evaluate the usability of Home Monitoring System for Heart Rate (BPM), in providing help to nurses, evaluating the overall clinical situation of post cardiac petients at home
To evaluate if Alerts and Flags generated by the EarlySense Home Care System, could have potentially prevented readmission to hospitals, and providing better care at home, for post cardiac surgery patients | 30 days
  Evaluate the usability of Home Monitoring System for Respiratory Rate (Br./min), in providing help to nurses, evaluating the overall clinical situation of post cardiac petients at home
To evaluate if Alerts and Flags generated by the EarlySense Home Care System, could have potentially prevented readmission to hospitals, and providing better care at home, for post cardiac surgery patients | 30 days
  Evaluate the usability of Home Monitoring System for activity indication such asnumber of bed exits during nighttime in providing help to nurses, evaluating the overall clinical situation of post cardiac petients at home
To evaluate if Alerts and Flags generated by the EarlySense Home Care System, could have potentially prevented readmission to hospitals, and providing better care at home, for post cardiac surgery patients | 30 days
  Evaluate the usability of Home Monitoring System activity indication such as number of hours spent in bed during the day in providing help to nurses, evaluating the overall clinical situation of post cardiac petients at home

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided